CLINICAL TRIAL: NCT04047667
Title: The Safety and Diagnostic Efficacy of Cone Beam CT Guided Transbronchial Cryobiopsy for ILD Patients
Brief Title: Cone Beam CT Guided Transbronchial Cryobiopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Dai Huaping, vice Director of Respiratory disease Center, China-Japan Friendship Hospital
Other Study IDs: ChinaJapanFH004
Record Dates: First submitted 2019-08-04; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: ILD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CBCT guided TBCB: Patients with ILD who met the following including criteria from September 2018 to July 2019 were suggested to receive TBCB under CBCT guidance: more than 18 years old, diffuse parenchymal lung diseases without a diagnosis after integration of clinical profile, laboratory tests and HRCT features, FVC more than 50%, DLCO more than 35%, patients without acute exacerbation within one month, patients without bleeding diathesis, anticoagulant therapy, using antiplatelet drugs, patients without pulmonary hypertension, respiratory failure, liver or kidney disfunction, or cardiac insufficiency, PLT more than 50 x 109/L. All included patients signed the informed consent.
  Interventions: Procedure: cone beam CT guided transbronchial cryobiopsy

INTERVENTIONS:
Procedure: cone beam CT guided transbronchial cryobiopsy — CBCT images are acquried and reviewed in axial, coronal and sagittal planes to most accurately assess the cryoprobe position within the lung parenchyma and relative to other thoracic structures. The minimum probe-to-pleura distance will be measured. If the position of cryoprobe is proper, TBCB will be perfomed.

SUMMARY:
Interstitial lung diseases (ILD) are common in clinical practices and need multidisciplinary assessment of clinical presentations, radiological and histological features. Transbronchial cryobiopsy (TBCB) is one of the most important invasive procedures for ILD when a confident diagnosis cannot be made by clinical and radiological assessment. TBCB could lead to higher incidence of risks. The pneumothorax and severe bleeding seemed to be more common in patients with TBCB.

Cone-beam computed tomography (CBCT) could provide 3-dimensinal (3D) CT images which were close to the image qualities of conventional CT. The probe-to-pleura relationship could be accurately established by the 3D CT scan and the cryobiopsy safety profile might be improved under the guidance of CBCT. In this study, we conducted a prospective study to observe the safety and diagnostic efficacy of CBCT guided TBCB for the DPLD patients.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old, diffuse parenchymal lung diseases without a diagnosis after integration of clinical profile, laboratory tests and HRCT features, FVC more than 50%, DLCO more than 35%

Exclusion Criteria:

* acute exacerbation within one month, bleeding diathesis, anticoagulant therapy, using antiplatelet drugs, patients with pulmonary hypertension, respiratory failure, liver, kidney disfunction, and cardiac insufficiency, PLT less than 50 x 109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ILD Patients without a diagnosis after integration of clinical profile, laboratory tests and HRCT features
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
safety profile of procedure | 30 days
  pneumothorax, bleeding severity, post-bronchoscopy fever, acute exacerbation of ILD, procedure related death.

SECONDARY OUTCOMES:
diagnostic efficacy | 30 days
  diagnostic yield

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bian Y, Deng M, Gao Q, Zhou G, Tong R, Zhao L, Liu M, Sun J, Dai H, Herth FJF, Hou G, Wang C. The Diagnostic Efficiency and Safety of Transbronchial Lung Cryobiopsy Using 1.1-mm Cryoprobe in Diagnosing Interstitial Lung Disease. Lung. 2024 Oct;202(5):615-623. doi: 10.1007/s00408-024-00713-2. Epub 2024 Jun 23. PMID 38910197
- [Derived] Bian Y, Zhou G, Gao Q, Deng M, Tong R, Xia Y, Lin J, Hou G, Dai H. Assessment of a randomized controlled trial on the safety of pre-placing bronchial balloons in transbronchial lung cryobiopsy for diagnosing interstitial lung disease. Eur J Med Res. 2024 May 3;29(1):268. doi: 10.1186/s40001-024-01871-y. PMID 38702744